CLINICAL TRIAL: NCT02897232
Title: Community and Physician Perspectives Regarding Male Youth Human Papillomavirus (HPV) Disease and Vaccination
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Julia M. Esparza, Head, User Education and Outreach Services, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: STUDY00000618
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Papillomavirus Infections; Health Behavior; Attitude of Health Personnel; Human Papilloma Virus, Male
Keywords: Human Papillomavirus Vaccine; HPV; Patient Acceptance; Physician Comfort; Male Vaccination; HPV Associated Cancers
MeSH Terms: conditions — Papillomavirus Infections; Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Community Group Survey: Community members coming into the University Health Shreveport Ambulatory Care Facility.
  Interventions: Other: Survey
- Physician Group Survey: Physicians affiliated with LSU Health Shreveport School of Medicine
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Clinical Faculty and community will be given a survey to define issues preventing HPV Vaccination

SUMMARY:
This is a minimal risk, anonymous, convenience sample, social behavioral study using qualitative descriptive survey methods. It is to ascertain community member, physician, resident and medical student perspectives regarding Human Papillomavirus (HPV) infection, associated diseases and to identify barriers which prevent these groups from ensuring that males 9-26 receive the three-shot vaccine series to prevent HPV infection.

The research is focused on these questions:

Do community members understand the ease of transmission of the HPV virus in males 9-26? Do community members, physicians, residents and medical students have knowledge of the associated diseases that may occur with the HPV virus infection in males age 9-26? Do community members, physicians, residents and medical students know the ages in which males should receive the HPV vaccine three-shot series? What barriers prevent community members and physicians, residents and medical students from ensuring that males 9-26 receive the three-shot vaccine series to prevent HPV infection?

DETAILED DESCRIPTION:
This is a minimal risk, anonymous, convenience sample, social behavioral study using qualitative descriptive survey methods. It is to ascertain community member, physician, resident and medical student perspectives regarding Human Papillomavirus (HPV) infection, associated diseases and to identify barriers which prevent these groups from ensuring that males 9-26 receive the three-shot vaccine series to prevent HPV infection.

The research is focused on these questions:

Do community members understand the ease of transmission of the HPV virus in males 9-26? Do community members, physicians, residents and medical students have knowledge of the associated diseases that may occur with the HPV virus infection in males age 9-26? Do community members, physicians, residents and medical students know the ages in which males should receive the HPV vaccine three-shot series? What barriers prevent community members and physicians, residents and medical students from ensuring that males 9-26 receive the three-shot vaccine series to prevent HPV infection?

ELIGIBILITY:
Community Participants

Inclusion

All visitors to the Pediatric or Internal Medicine University Health Shreveport Clinics willing to complete a survey

Community Study Exclusion

Those do not wish to participate in the study

Those who English is not their first language

Clinical Faculty, Resident, and Medical Student Study

Inclusion

All Louisiana State University Shreveport Health Clinical Faculty, Resident, and Medical Student Inclusion willing to to complete the online survey.

Clinical Faculty, Resident, and Medical Student Study

Exclusion

Any LSU Health Shreveport Clinical Faculty, Resident, and Medical Student which declines to take the survey or do not attempt to complete it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Northern Louisiana community members in the Ambulatory Care Clinics in University Health.
  Northern Louisiana, Louisiana State University Health, clinical faculty, residents and medical students.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Barriers to HPV Vaccination | 60 days
  What are the barriers which prevent community members and physicians, residents and medical students from ensuring that males age 9-26 are vaccinated with the HPV three-shot vaccination.

SECONDARY OUTCOMES:
Knowledge pertaining to ease of Human Papillomavirus transmission. | 60 days
  Do community members and physicians understand the ease of HPV transmission?
Knowledge of Associated HPV diseases | 60 days
  Do community member and physicians know the associated HPV diseases?
Knowledge of age in which males should be vaccinated against HPV. | 60 days
  Do community member and physicians know the age in which males should be vaccinated against HPV?

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Esparza, MLS, Principal Investigator — 3186754179
Locations (1):
- Louisiana State University Health, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.